CLINICAL TRIAL: NCT02481726
Title: 68Ga-AlfatideII for the Differential Diagnosis of of Lung Cancer and Lung Tuberculosis by PET/CT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: XijingH
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Lung Cancer; Lung Tuberculosis
Keywords: 68Ga; Alfatide II; RGD; αvβ3; PET/CT
MeSH Terms: conditions — Lung Neoplasms; Tuberculosis, Pulmonary | interventions — alfatide II; Fluorodeoxyglucose F18

ARMS (1):
- 68Ga (Experimental): In patients in suspicion of lung cancer or lung tuberculosis; in patients with differential diagnosis difficulties; without treatment or surgery. They underwent a standard routine 18F-FDG PET/CT first, and were injected 10~20MBq 68Ga-Alfatide II in the next day, followed by whole body PET/CT acquisitions.
  Interventions: Radiation: 68Ga-labeled peptides of dimer RGD (Alfatide II) and 18F-FDG

INTERVENTIONS:
Radiation: 68Ga-labeled peptides of dimer RGD (Alfatide II) and 18F-FDG

SUMMARY:
Comparison of 68Ga-AlfatideII and 18F-FDG in differential diagnosis effectiveness towards the solitary pulmonary nodules of lung cancer or tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide a written informed consent
* Males and females, ≥18 years old.
* The definite diagnosis of lung cancer was established by pre-operational bronchoscopic or puncture biopsy or the definite diagnosis of lung tuberculomas was established on the basis of positive sputum culture examinations and confirmed by follow-up.
* Without any treatment or resection surgury.
* All the biopsies are done at least 10 days before PET/CT scans.
* Evaluation of cardiac function.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential；
* Known severe allergy or hypersensitivity to IV radiographic contrast；
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the investigator, may significantly interfere with study compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Quantitative measurement of standardized uptake values (SUVs) of lesions. | 1 year
  The quantitative analysis will be performed by the same person for all cases, and the standardized uptake value (SUV) of each tumor will be measured using a volume of interest (VOI) method.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety after 68Ga-NEB injection and PET/CT scanning. | 1 year